CLINICAL TRIAL: NCT06055127
Title: Osseodensifiction Versus Piezoelectric Internal Sinus Elevation (PISE) Technique in Delayed Implant Placement (A Randomized Controlled Clinical Trial)
Brief Title: Osseodensifiction Versus Piezoelectric Internal Sinus Elevation Technique in Delayed Implant Placement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohammed Samir, Resident ( Principal Investigator), Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FDASU_Rec IM 122215
Record Dates: First submitted 2023-09-16; First posted 2023-09-26 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Maxillary Sinus Floor Augmentation
Keywords: internal sinus elevation; osseodensfication,; piezoelectric surgery

STUDY DESIGN:
Intervention Model Description: parallel single blind masking randomized controlled clinical trail
Who Masked: Participant
Masking Description: computer-generated randomization table
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- osseodensifiction internal sinus lift / sticky bone graft material (Experimental): Osseodensifiction compacts bone and simultaneously autografts it into the osteotomy walls and apex instead of removing it. The use of a Densah® drill bit at high speed counterclockwise, without a cutting edge and with a steady irrigation causes the formation of a layer of strong dense bone along the walls of the base of the osteotomy preparation.
  Interventions: Procedure: osseodensifiction internal sinus lift / sticky bone graft material
- piezoelectric internal sinus lift / sticky bone graft material (Active Comparator): The piezoelectric surgical sets comprise various inserts from osteotomies to diamond-cutting inserts. The hydropneumatics pressure of the saline solution irrigation is subjected to the piezoelectric cavitation pushing the Schneiderian membrane upwards resulting in its' detachment and floating
  Interventions: Procedure: piezoelectric internal sinus lift / sticky bone graft material

INTERVENTIONS:
Procedure: osseodensifiction internal sinus lift / sticky bone graft material — The osteotomy for the osseodensification internal sinus lift begins with a twist drill advanced at 800 rpm with saline irrigation to within 1-2 mm from the sinus floor. Next, a series of osteotomy drills are used in the same fashion at 800 rpm to widen the osteotomy. The final osteotomy drill is advanced with gentle pressure at 100 rpm counterclockwise without irrigation until a bouncing sensation occurs "haptic feedback" at this point infracture of the sinus has taken place. After infracture, injection of the graft material into the osteotomy site will occur. The final osteotomy drill is used to guide the graft apically. This process is repeated in an incremental fashion to lift the membrane. Once enough space has been created below the antral membrane, implant insertion will occur then suturing.
  Arms: osseodensifiction internal sinus lift / sticky bone graft material
Procedure: piezoelectric internal sinus lift / sticky bone graft material — In the PISE technique, an ultrasonic piezoelectric device (acteon), to which a specialized tip is attached, is used to break the sinus floor. Developed for sinus lift by the crestal approach, the Intralift™ Kit makes it possible to undertake dental non invasive surgery in full safety.
  The diamond-coated tips, of increasing diameters (from 1.35mm to 2.80mm), are designed to drill and gradually widen the access canal to the sinus membrane. The sterile spray cools the tips down to avoid any rise in temperature, which could lead to oral tissue damage.The membrane elevation is achieved using the TKW5 by means of microcavitation. Thanks to the ultrasonic frequency modulation, the risk of membrane damage is limited. Moreover, the cavitation effect enables excellent visibility of the operating field.
  Arms: piezoelectric internal sinus lift / sticky bone graft material

SUMMARY:
The present study is a parallel single-blinded randomized controlled clinical trial.

The study will be conducted after being reviewed and approved by the Faculty of Dentistry, AinShams University Research Ethics Committee (FDASU-REC).

The study population will be randomly allocated into two groups of the same size:

Group 1: Osseodensifiction sinus lift will be performed using sticky bone as a graft material.

Group 2: Piezoelectric Internal Sinus Elevation (PISE) will be performed using sticky bone as a graft material.

The aim of the present study is to evaluate the effectiveness and clinical results of osseodensification in comparison to Piezoelectric Internal Sinus Elevation (PISE) Technique in Delayed Implant Placement.

ELIGIBILITY:
Inclusion Criteria:

1. Patient partially edentulous with maxillary posterior edentulous ridge after extraction of more than 4 months.
2. Both sexes will be selected males and females.
3. Adult patients aged between 18 and 40 years of age.
4. Good general health (American Society of Anesthesiology Physical Status Ⅰ-Ⅱ).
5. Initial residual alveolar ridge height ranging between 4 to 6 mm according to preoperative CBCT.
6. No previous surgery or radiation treatment on the maxillary sinus.

Exclusion Criteria:

* 1. Smokers. 2. Pregnant or lactating females. 3. Psychiatric disorders. 4. Uncontrolled systemic disease. 5. Hematologic diseases and coagulation disorders. 6. Chemotherapy or radiotherapy of the head and neck area, and immunocompromised status.

  7. Medical conditions affecting bone metabolism and ongoing treatment with bisphosphonates drugs or systemic steroids.

  8. Presence of acute or chronic sinus pathoses or sinus membrane perforation.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2023-09-08 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Radiographic assessment of change in the vertical bone height (bone gain) | per-operative and immediately post-operative
  Immediate postoperative CBCTs will be taken to all participants to assess bone gain .
Radiographic assessment of bone density | per-operative and immediately post-operative
  Immediate postoperative CBCTs will be taken to all participants to assess bone density.

SECONDARY OUTCOMES:
implant primary stability (insertion torque ) | during procedure
  implant insertion torque will be assessed using torque wrench .
implant primary stability (ISQ) | during procedure
  implant stability quotient will be assessed using Osstell device
patient post-operative pain assessment | 1 week post-operative
  obtained using a 100 mm visual analogue scale
patient's satisfaction assessment | 1 week post-operative
  obtained by the aid of a health-related quality of life questionnaire
operator's satisfaction assessment | 1 year
  obtained by the aid of a questionnaire assessing the operator's satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Samir, BDs, Principal Investigator — AinShams University
Locations (1):
- AinShams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huwais S, Mazor Z, Ioannou AL, Gluckman H, Neiva R. A Multicenter Retrospective Clinical Study with Up-to-5-Year Follow-up Utilizing a Method that Enhances Bone Density and Allows for Transcrestal Sinus Augmentation Through Compaction Grafting. Int J Oral Maxillofac Implants. 2018 Nov/Dec;33(6):1305-1311. doi: 10.11607/jomi.6770. PMID 30427961
- [Background] Pjetursson BE, Lang NP. Sinus floor elevation utilizing the transalveolar approach. Periodontol 2000. 2014 Oct;66(1):59-71. doi: 10.1111/prd.12043. PMID 25123761
- [Background] Torrella F, Pitarch J, Cabanes G, Anitua E. Ultrasonic ostectomy for the surgical approach of the maxillary sinus: a technical note. Int J Oral Maxillofac Implants. 1998 Sep-Oct;13(5):697-700. PMID 9796155
- [Background] Li J, Lee K, Chen H, Ou G. Piezoelectric surgery in maxillary sinus floor elevation with hydraulic pressure for xenograft and simultaneous implant placement. J Prosthet Dent. 2013 Nov;110(5):344-8. doi: 10.1016/j.prosdent.2013.04.002. Epub 2013 Sep 29. PMID 24084145
- [Background] Mourao CF, Valiense H, Melo ER, Mourao NB, Maia MD. Obtention of injectable platelets rich-fibrin (i-PRF) and its polymerization with bone graft: technical note. Rev Col Bras Cir. 2015 Nov-Dec;42(6):421-3. doi: 10.1590/0100-69912015006013. English, Portuguese. PMID 26814997
- [Derived] Samir M, Bissar MW, Abuel-Ela HA. Osseodensification versus piezoelectric internal sinus elevation (PISE) technique in delayed implant placement (a randomized controlled clinical trial). BMC Oral Health. 2024 Oct 28;24(1):1306. doi: 10.1186/s12903-024-04964-6. PMID 39468538